CLINICAL TRIAL: NCT06424301
Title: Targeting NUDT21 siRNA Drugs for Patients With Refractory Retinoblastoma (A Prospective Pilot Study)
Brief Title: Targeting NUDT21 siRNA Drugs for Patients With Refractory Retinoblastoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Collaborators: The Eye Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDEENT-20241031
Record Dates: First submitted 2024-05-16; First posted 2024-05-22 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Retinoblastoma; Refractory
Keywords: retinoblastoma; intravitreal Chemotherapy
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravitreal chemotherapy in patients with refractory retinoblastoma (Experimental): Prior to the first administration of the targeted drug, enrolled patients underwent peripheral blood sampling and comprehensive clinical evaluation. Intravitreal injections of the targeted drug were administered at a dosage of 100-200 μg (100 μg for patients under 2 years of age; 200 μg for patients aged 2 years and above) on Day 1 of Weeks 1, 3, and 7. Aqueous humor samples were collected at the time of injection during Weeks 1, 3, and 7. Clinical assessments were conducted monthly, with continuous follow-up extending through Week 24.
  Interventions: Drug: Targeting NUDT21 siRNA drugs

INTERVENTIONS:
Drug: Targeting NUDT21 siRNA drugs — It is performed for intravitreal chemotherapy.

SUMMARY:
Retinoblastoma (RB) is the most common intraocular malignancy in children, accounting for approximately 11% of all cancers diagnosed in children under the age of one. Although its incidence is relatively low-about 1 in 15,000 to 20,000 live births-RB has a high risk of intracranial metastasis via the optic nerve, often leading to poor prognosis in advanced cases.

Recent advances in administration routes, such as intravitreal and intra-arterial chemotherapy, have significantly improved eye preservation rates. However, these strategies are limited by cumulative retinal toxicity and drug resistance. In refractory cases, enucleation remains the only definitive treatment to prevent extraocular spread and death.

In light of these challenges, current research efforts are focused on developing novel targeted therapies that enhance anti-tumor efficacy while minimizing local toxicity. In this context, we introduce a first-in-class siRNA-based drug targeting NUDT21, which promotes tumor regression by modulating the 3'UTR tail of SMC1A, thereby suppressing tumor cell proliferation. Importantly, the siRNA drug selectively targets tumor cells, offering a favorable safety profile compared to conventional chemotherapeutic regimens.

Given that both the target (NUDT21) and the mode of administration (intraocular siRNA injection) are novel in retinoblastoma treatment, there is an urgent need for early-phase investigator-initiated clinical research. This study is therefore designed to assess the short-term safety and preliminary efficacy of NUDT21 siRNA in patients with refractory retinoblastoma, and to provide an evidence base for future large-scale clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with retinoblastoma with a somatic mutation of the gene RB1 and active tumor in a single eye, or germinal mutation of RB1 with active tumor/s in an eye and the contralateral eye unaffected, enucleated or without tumor activity. In both cases, relapsed or refractory with the use of systemic, intraarterial or intravitreal chemotherapy or radiotherapy, in accordance with the availability at his/her referral site, in whom enucleation is the only recommended treatment under opinion of the medical team treating the case at the originating referral site. But the patient has a strong desire to preserve the eye.
2. Normal renal function: serum creatinine: < 45 μmol/L (0-2 years); < 57 μmol/L (3-6 years); < 60 μmol/L (7-10 years); < 80 μmol/L (11-13 years).
3. Normal Hepatic function: serum ALT: < 0,52 μkat/L (de 9 months -12 years); serum AST: 61-80 g/L (8 months - 5 years); 63-83 g/L (5-9 years); 63-82 g/L (9-12 years).
4. Age greater than 6 months at the time of inclusion in the study.
5. Sign the informed consent form and be willing to follow up at the specified time.

Exclusion Criteria:

1. Presence of factors that require immediate enucleation of the affected eye such as glaucoma, rubeosis iridis, anterior chamber involvement.
2. Comorbidities: Uncontrolled epilepsy with anticonvulsant treatment, cardiac disease not compensated by treatment.
3. Active Infections.
4. Other chronic or active acute diseases that under the criterion of the researcher were an exclusion criterion.
5. History of having received attenuated or live vaccines in the 30 days prior to inclusion in the study.
6. Any cause of Immunosuppression.
7. Trilateral Retinoblastoma.
8. Extraocular spread.
9. History of having received treatment for retinoblastoma with chemotherapy or radiation therapy by any means within 30 days prior to inclusion in the study.
10. Patients who can not complete the study procedures.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-12-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 months
  Treatment-emergent adverse events (TEAEs) are defined as any unfavorable or unintended sign, symptom, or disease temporally associated with the administration of intravitreal siRNA therapy, whether or not considered related to the drug. Use CTCAE v5.0 (Common Terminology Criteria for Adverse Events) for grading severity.

SECONDARY OUTCOMES:
Tumor size | 6 months
  Tumor size will be assessed by measuring tumor thickness (height) from the retinal surface to the apex of the lesion on optical coherence tomography (OCT) scan. Serial OCT scans will be used to track tumor regression or progression over time. This outcome aims to assess anatomical response to treatment and provide imaging-based evidence of therapeutic efficacy.
Retinal function | 6 months
  Photopic flicker electroretinography (ERG) will be conducted in accordance with ISCEV standards, typically using a 30 Hz stimulus. The amplitude will be measured and compared pre- and post-treatment. This outcome will assess the potential impact of the investigational therapy on cone system integrity and retinal functional preservation.
Target engagement | 6 months
  We will measure the concentrations of NUDT21 and SMC1A proteins in aqueous humor samples using enzyme-linked immunosorbent assay (ELISA) before and after treatment. This assessment will confirm pharmacodynamic target engagement of the NUDT21 siRNA therapy by evaluating changes in NUDT21 and downstream effector SMC1A expression levels.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Zhao, MD, Principal Investigator — Fudan Eye & ENT Hospital; Kang Xue, MD, Study Director — Fudan Eye & ENT Hospital; Kang Zhang, MD, Study Director — The Eye Hospital of Wenzhou Medical University; Jiang Qian, MD, Study Director — Fudan Eye & ENT Hospital
Locations (1):
- Fudan Eye & ENT Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared upon requirement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code